CLINICAL TRIAL: NCT02759770
Title: Risk Factors and Prediction Score of ARDS After Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Guangfa Zhu, chief physician, Beijing Anzhen Hospital
Other Study IDs: Shoufa-2016-2-1052
Record Dates: First submitted 2016-04-25; First posted 2016-05-03 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2019-12

CONDITIONS: Respiratory Distress Syndrome, Adult; Thoracic Surgery; Risk Factors
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (3):
- ARDS: ARDS patients after cardiac surgery
  Interventions: Other: no intervention
- non-ARDS: non-ARDS patients after cardiac surgery
  Interventions: Other: no intervention
- propective group: patients of cardiac surgery including ARDS and non-ARDS patients
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is a clinical observational study, no intervention was included.

SUMMARY:
Acute respiratory distress syndrome following cardiac surgery severely affects the prognosis of patients; the mortality is up to 40%. Although experience many years of research and exploration, the effective methods for the treatment of acute respiratory distress syndrome is still relatively limited at present, including lung protective mechanical ventilation respiratory support, fluid management, glucocorticoid and other integrated organ function maintenance measures. It is currently the research of acute respiratory distress syndrome aims at the early discovery and takes effective measures to prevent its occurrence, hoping to improve the prognosis of patients. According to risk factors is established through the analysis of lung injury score early warning system, the early identification of acute respiratory distress syndrome patients at high risk, before the occurrence of acute respiratory distress syndrome take corresponding preventive measures can effectively reduce the incidence rate and mortality. So far, domestic and foreign research on the establishment of acute respiratory distress syndrome scoring early warning system is less. Cardiac surgery has significant characteristics, type of operation, location, operation, intraoperative blood transfusion and oxygenation, postoperative factors, are likely to be the factors of acute respiratory distress syndrome. As far as investigators know, so far there are few specialized for acute respiratory distress syndrome predicting lung injury after cardiac surgery. This study will be completed after the implementation of individualized dynamic lung injury score evaluation of cardiac surgery patients, identification of high-risk acute respiratory distress syndrome patients, to assist clinicians in early decision, take preventive measures. This study will improve the prognosis of acute respiratory distress syndrome patients after cardiac surgery; it is of great significance to improve the level of intensive care after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Retrospective group: cardiac surgery patients accepted from Jan 2013 to Dec 2015
* Prospective group: cardiac surgery patients accepted from 2017 January to December

Exclusion Criteria:

* refused to participate in the study
* age less than 18 years old
* before operation performed mechanical ventilation
* before operation underwent IABP treatment
* before operation continuous renal replacement therapy
* before operation undergoing in vitro membrane oxygenator treatment
* before operation has the pulmonary imaging showed bilateral pulmonary diffuse exudation of interstitial pneumonia, pulmonary infection or respiratory failure
* the major trauma, sepsis, aspiration, shock, acute heart failure
* before operation diagnosed as malignant tumor
* Incomplete data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of cardiac surgery in Beijing Anzhen hospital
Sampling Method: Non-Probability Sample
Enrollment: 1333 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
The number of acute respiratory distress syndrome following cardiac surgery in Anzhen hospital during Jan 2013 to Dec 2015. | up to 12months
The number of patients of cardiac surgery in Anzhen hospital during Jan 2013 to Dec 2015. | up to 12months
The number of acute respiratory distress syndrome following cardiac surgery in Anzhen hospital during Jan 2017 to Dec 2017. | up to 12months
The number of patients of cardiac surgery in Anzhen hospital during Jan 2017 to Dec 2017. | up to 12months
The number of diabetic patients in ARDS group. | up to 1 month
The number of diabetic patients in non-ARDS group. | up to 1 month
The number of chronic obstructive pulmonary disease patients in ARDS group. | up to 1 month
The number of chronic obstructive pulmonary disease patients in non-ARDS group. | up to 1 month
The type of operation in ARDS group. | up to 1 month
The type of operation in non-ARDS group. | up to 1 month
The body mass index in ARDS group. | up to 1 month
The body mass index in non-ARDS group. | up to 1 month
The heart function in ARDS group before operation. | up to 1 month
The heart function in non-ARDS group before operation. | up to 1 month
The oxygenation in ARDS group before operation. | up to 1 month
The oxygenation in non-ARDS group before operation. | up to 1 month
The drug taken by patients in ARDS group. | up to 1 month
The drug taken by patients in non-ARDS group. | up to 1 month
The nutrition situation of patients in ARDS group. | up to 1 month
The nutrition situation of patients in non-ARDS group. | up to 1 month
The process of operation in ARDS group. | up to 1 month
The process of operation in non-ARDS group. | up to 1 month
The blood transfusion of patients during operation in ARDS group. | up to 1 month
The blood transfusion of patients during operation in non-ARDS group. | up to 1 month
The oxygenation of patients during operation in ARDS group. | up to 1 month
The oxygenation of patients during operation in non-ARDS group. | up to 1 month
The drug taken by patients after operation in ARDS group. | up to 1 month
The drug taken by patients after operation in non-ARDS group. | up to 1 month
The oxygenation of patients after operation in ARDS group. | up to 1 month
The oxygenation of patients after operation in non-ARDS group. | up to 1 month
The situation of mechanical ventilation of patients after operation in ARDS group. | up to 1 month
The situation of mechanical ventilation of patients after operation in non-ARDS group. | up to 1 month

SECONDARY OUTCOMES:
The mortality of acute respiratory distress syndrome following cardiac surgery in Anzhen hospital . | up to 1months
The morbidity of acute respiratory distress syndrome following cardiac surgery in Anzhen hospital . | up to 1months

CONTACTS AND LOCATIONS:
Overall Officials: Guangfa Zhu, Study Chair — Department of Respiratory and Critical Care Medicine, Beijing Anzhen Hospital, Capital Medical University, Beijing Institute of Heart, Lung and Blood Vessel Diseases
Locations (1):
- Department of Respiratory and Critical Care Medicine, Beijing Anzhen Hospital, Capital Medical University, Beijing Institute of Heart, Lung and Blood Vessel Diseases, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Kogan A, Preisman S, Levin S, Raanani E, Sternik L. Adult respiratory distress syndrome following cardiac surgery. J Card Surg. 2014 Jan;29(1):41-6. doi: 10.1111/jocs.12264. Epub 2013 Dec 3. PMID 24299028
- [Background] Berg KS, Stenseth R, Pleym H, Wahba A, Videm V. Mortality risk prediction in cardiac surgery: comparing a novel model with the EuroSCORE. Acta Anaesthesiol Scand. 2011 Mar;55(3):313-21. doi: 10.1111/j.1399-6576.2010.02393.x. PMID 21288212
- [Background] Forel JM, Voillet F, Pulina D, Gacouin A, Perrin G, Barrau K, Jaber S, Arnal JM, Fathallah M, Auquier P, Roch A, Azoulay E, Papazian L. Ventilator-associated pneumonia and ICU mortality in severe ARDS patients ventilated according to a lung-protective strategy. Crit Care. 2012 Dec 12;16(2):R65. doi: 10.1186/cc11312. PMID 22524447
- [Background] Grissom CK, Hirshberg EL, Dickerson JB, Brown SM, Lanspa MJ, Liu KD, Schoenfeld D, Tidswell M, Hite RD, Rock P, Miller RR 3rd, Morris AH; National Heart Lung and Blood Institute Acute Respiratory Distress Syndrome Clinical Trials Network. Fluid management with a simplified conservative protocol for the acute respiratory distress syndrome*. Crit Care Med. 2015 Feb;43(2):288-95. doi: 10.1097/CCM.0000000000000715. PMID 25599463
- [Background] Festic E, Kor DJ, Gajic O. Prevention of acute respiratory distress syndrome. Curr Opin Crit Care. 2015 Feb;21(1):82-90. doi: 10.1097/MCC.0000000000000174. PMID 25501020
- [Background] Rubenfeld GD. Who cares about preventing acute respiratory distress syndrome? Am J Respir Crit Care Med. 2015 Feb 1;191(3):255-60. doi: 10.1164/rccm.201408-1574CP. PMID 25478722
- [Background] Beitler JR, Schoenfeld DA, Thompson BT. Preventing ARDS: progress, promise, and pitfalls. Chest. 2014 Oct;146(4):1102-1113. doi: 10.1378/chest.14-0555. PMID 25288000
- [Background] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452
- [Background] Milot J, Perron J, Lacasse Y, Letourneau L, Cartier PC, Maltais F. Incidence and predictors of ARDS after cardiac surgery. Chest. 2001 Mar;119(3):884-8. doi: 10.1378/chest.119.3.884. PMID 11243972
- [Background] Michalopoulos A, Prapas S, Falagas ME. The incidence of adult respiratory distress syndrome in patients undergoing off-pump coronary artery bypass grafting surgery. Eur J Anaesthesiol. 2006 Jan;23(1):80. doi: 10.1017/S0265021505211821. No abstract available. PMID 16390572
- [Background] Vakili M, Shirani S, Paknejad O, Yousefshahi F. Acute Respiratory Distress Syndrome diagnosis after coronary artery bypass: comparison between diagnostic criteria and clinical picture. Acta Med Iran. 2015;53(1):51-6. PMID 25597606
- [Background] Kor DJ, Lingineni RK, Gajic O, Park PK, Blum JM, Hou PC, Hoth JJ, Anderson HL 3rd, Bajwa EK, Bartz RR, Adesanya A, Festic E, Gong MN, Carter RE, Talmor DS. Predicting risk of postoperative lung injury in high-risk surgical patients: a multicenter cohort study. Anesthesiology. 2014 May;120(5):1168-81. doi: 10.1097/ALN.0000000000000216. PMID 24755786